CLINICAL TRIAL: NCT00651716
Title: Regulatory T Cells at Engraftment as Predictors of Acute Graft-Versus-Host Disease Outcomes in Patients Undergoing Allogeneic Stem Cell Transplantation
Brief Title: T Cells in Predicting Acute Graft-Versus-Host Disease in Patients Undergoing Donor Stem Cell Transplant
Status: Terminated | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Brian Engelhardt, MD, Assistant Professor of Medicine; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BMT 0653; P30CA068485 (NIH)
Record Dates: First submitted 2008-04-02; First posted 2008-04-03 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Carcinoma, Ovarian Epithelial; Testicular Neoplasms | interventions — Flow Cytometry; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allogeneic Stem Cell Transplant Patients: Patients undergoing allogeneic stem cell transplant (SCT). Potential study candidates will be identified by participating physicians.
  Interventions: Other: flow cytometry; Other: laboratory biomarker analysis; Other: Data Collection

INTERVENTIONS:
Other: flow cytometry — Lymphocyte Analysis: Lymphocyte subset studies will be performed on samples obtained from the patient, donor, or graft. Aliquots will be analyzed using standard flow cytometry.
Other: laboratory biomarker analysis — Identification of gut-homing and skin-homing Treg subsets
Other: Data Collection — Patient samples will receive an alphanumeric code assigned by the principal investigator so that patient and donor identity will be known only to study investigators and research staff. Clinical records on each patient will be reviewed by participating investigators or research staff on a routine basis so that relevant clinical information including survival, malignancy relapse, and GVHD can be included in the patient database. Flow cytometry results will also be included in this database.

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors predict whether patients undergoing donor stem cell transplant will develop acute graft-versus-host disease.

PURPOSE: This clinical trial is studying T cells to see how well they help in predicting acute graft-versus-host disease in patients undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the association between regulatory T-lymphocyte (Treg) subsets present at engraftment and at day 28 with the incidence of acute graft-versus-host-disease (aGVHD) in patients undergoing allogeneic stem cell transplantation.
* To identify gut-homing and skin-homing Treg subsets and determine their role during engraftment and at day 28 as a predictor of gut and skin aGVHD, respectively.

OUTLINE: Patients undergo blood sample collection at the time of neutrophil engraftment prior to stem cell transplant (SCT) and post-SCT on days 7, 14, 21, and 28 days after allogeneic stem cell transplantation. Blood samples are analyzed for T-cell subsets and for the percentage of regulatory T-lymphocyte (Treg) or other T-cell subsets expressing specific homing receptors for the gut or skin via flow cytometry.

Patients' medical records are also reviewed periodically.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing allogeneic SCT
* Age >= 18 years

Exclusion criteria:

* Inability to give informed consent
* Patients who have not received an allogeneic SCT
* Any condition which, in the opinion of the investigator, might interfere with study objective
* Any reason which, in the opinion of the investigator, adds additional risk to the patient

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a disease which is being treated with a bone marrow and/or a stem cell transplant.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Percentage of regulatory T-lymphocytes (Tregs) at engraftment | day of stem cell transplant
  percentage of Treg subsets present in patient's blood before they undergo stem cell transplant

SECONDARY OUTCOMES:
Association between Treg subsets and acute graft-vs.-host disease outcomes | at stem cell transplant and at day 28
  Identify gut homing and skin homing Treg lymphocyte subsets and compare and contrast them to determine links between the Treg subsets and gut and/or skin acute graft-vs.-host-disease incidence, stage/grade, target organ involvement, and responsiveness to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Engelhardt, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/